CLINICAL TRIAL: NCT02954705
Title: MICRO-RNAs OF NEUTROPHILS IN RENAL ANCA-ASSOCIATED VASCULITIS
Brief Title: MICRO-RNAs OF NEUTROPHILS IN RENAL ANTINEUTROPHIL CYTOPLASMIS ANTIBODY (ANCA) -ASSOCIATED VASCULITIS
Acronym: MINERVA
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: RC15_0454
Record Dates: First submitted 2016-11-02; First posted 2016-11-03 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: ANCA-associated Vasculitis
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 50 mL of blood and 10 mL of urine by patient
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group AAV: Patients recruited from the Nantes University Hospital. 50 milliliter of blood and 10mL of urine are collected from these patients during levies in clinical visit.
  Interventions: Other: Non interventional study
- Group control: People recruited from the "Etablissement français du sang" (French blood establishment ).
  10 milliliter of blood are collected from these donors
  Interventions: Other: Non interventional study

INTERVENTIONS:
Other: Non interventional study — This is a non interventional study because all levies are performed during visit planned for the care of patients.

SUMMARY:
Activation of neutrophils by ANCA ("Anti-Neutrophil Cytoplasm Antibodies") and subsequent microvascular endothelial cell damage is the main feature of ANCA-associated vasculitis (AAV), a severe autoimmune disease that often targets the kidney. There is no specific treatment for AAV to date and 25% of patients with renal damage evolve towards end-stage renal disease, requiring dialysis and kidney transplantation. In addition, there is no reliable biological marker of the disease activity available, which makes the diagnostic, follow-up and treatment of patients difficult. Therefore, the identification of new therapeutic targets and non-invasive biomarkers constitutes a major clinical challenge to improve AAV patients care and to ameliorate their renal outcome.

ELIGIBILITY:
Inclusion Criteria for patients:

* Adult patients aged over 18 years
* Patients with Granulomatosis with polyangiitis or microscopic polyangiitis meeting the criteria of Chapel Hill.
* corticosteroid treatment <20 mg / day.
* Informed consent: oral for participation in research and writing for biological collection.

Inclusion Criteria for controls patients:

- healthy-topics matched for age, recruited from the Etablissement français du sang or in the Department of Internal Medicine of Nantes University Hospital

Non Inclusion Criteria:

* ANCA-associated vasculitis with Eosinophilic granulomatosis with polyangiitis (AAV-EGPA).
* Infectious or progressive tumor pathology.
* Pregnancy, lactation
* Treatment with cyclophosphamide in the 6 months prior to inclusion.
* Terminal chronic renal failure, presence of organ allograft.
* Thrust Patients receiving corticosteroids> 20 mg / d in the previous 4 weeks.
* Inability to give informed about information (subject in emergencies, understanding of the subject of difficulty, ...)
* Minor subject, under judicial protection, guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This will be done in total in 50 patients with ANCA-associated vasculitis (AAV) and 20 control patients. Among the 50 patients with AAV, 30 patients will be newly diagnosed and 20 already followed for AAV
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Expression profile of miRNAs in patients with AAV in circulating neutrophils, plasma and urine. | 6 month after maintenance treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fadi Fakhouri, Pr, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No